CLINICAL TRIAL: NCT06331845
Title: Stop and go Strategy as First-line Treatment in Patients With Objective Response After Systematic Chemotherapy for Widely de Novo Metastatic Nasopharyngeal Carcinoma: A Phase II Trial
Brief Title: Stop and go Strategy as First-line Treatment for Widely Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC012
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Intermittent Systematic Chemotherapy
Keywords: metastatic nasopharyngeal carcinoma; systematic chemotherapy; intermittent systematic chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Taxes; Capecitabine; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intermittent systematic chemotherapy group (Experimental): Patients diagnosed with wmNPC (more than five metastatic lesions) by histopathology are assigned to receive ISC following SC. Typically, SC(GP) was administered once every three weeks, with a maximum of six courses. Following this, ISC (TS1) was administered to extend the chemotherapy interval, once every 6-8 weeks, until widely progressive disease (WPD: defined as more than five progressive lesions), treatment intolerance, or patient refusal.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Paclitaxel protein-bound; Drug: Capecitabine; Drug: Tislelizumab

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 on Days 1 and 8
Drug: Cisplatin — a total of 80-100 mg/m2 for d1-3
Drug: Paclitaxel protein-bound — 260 mg/m2 on Day 1
Drug: Capecitabine — a dose of 1-1.25 g/m2 twice daily in in 2 weeks for one cycle
Drug: Tislelizumab — 200 mg on Day 1

SUMMARY:
This study aimed to investigate the value of a novel strategy of intermittent systematic chemotherapy (ISC) in widely metastatic nasopharyngeal carcinoma (wmNPC) patients who achieve objective response after systematic chemotherapy (SC).

DETAILED DESCRIPTION:
Widely metastatic nasopharyngeal carcinoma (wmNPC) represented a particular subgroup of patients with the worst prognosis, of which palliative systematic chemotherapy(SC) was recommended as initial treatment, however, palliative systematic treatment was often required to be stopped due to the cumulative toxicities while stopping SC may lead to disease progression, a 'stop and go' approach, namely chemotherapy 'holidays', was a new strategy which may keep a good balance of benefit and risk. This study aimed to investigate the value of a novel strategy of intermittent systematic chemotherapy (ISC) in wmNPC patients who achieve objective response after SC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple metastases at first diagnosis or multiple metastases after treatment(multiple metastases were defined as more than 5 lesions and/or more than 2 metastasis organs); Histologically or cytologically confirmed multiple metastatic NPC.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at trial entry, and life expectancy ≥ 6 months as judged by the Investigator;
3. The disease must be measurable with at least 1 unidimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; Adequate organ function;
4. Take adequate contraceptive measures throughout the study, and contraception continues until 12 months after treatment;
5. Able and willing to provide a signed informed consent form, and able to comply with all procedures.
6. The time from the last chemotherapy and/or radiotherapy to randomization must be ≥6 months.

Exclusion Criteria:

1. Patients with a hypersensitivity to any of the drugs used in our study;
2. With any active autoimmune disease or history of autoimmune disease;
3. Clinically significant cardiovascular and cerebrovascular diseases;
4. Have or are suffering from other malignant tumors within 5 years (except non-melanoma skin cancer or pre-invasive cervical cancer);
5. Active systemic infection;
6. Drug or alcohol abuse;
7. No or limited capacity for civil conduct;
8. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
9. History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy；
10. Use cortisol or other systematic immunosuppressive medications within 4 weeks before the study treatment, and the subject requiring hormone therapy during trials.
11. Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 1 year
  the time interval from the start of chemotherapy to the date of progression

SECONDARY OUTCOMES:
progression-free survival 2 | 1 year
  the time interval from the start of chemotherapy to the date of wide progression
overall survival | 1 year
  time from the date of the start of chemotherapy to death due to any cause